CLINICAL TRIAL: NCT03361956
Title: A Phase 2a, Randomized, Partially-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Pharmacokinetics of Treatment With Multiple Doses of JNJ-56136379 as Monotherapy and in Combination With a Nucleos(t)Ide Analog in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: An Efficacy, Safety, and Pharmacokinetics Study of JNJ-56136379 in Participants With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108410; 2017-001110-29 (EudraCT Number); 56136379HPB2001 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — JNJ-56136379; Sodium; entecavir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A: Arm 1 (JNJ-56136379 or NA) (open label) (Experimental): Participants with hepatitis B virus (HBV) currently not being treated and receiving JNJ-56136379 tablet (at a lower dose) orally for 24 weeks, will stop further dosing with JNJ-56136379 and start treatment with nucleos(t)ide analog (NA) (entecavir [ETV] or tenofovir disoproxil fumarate [TDF]), and enter the 24 week post treatment follow-up phase.
  Interventions: Drug: JNJ-56136379; Drug: NA (ETV or TDF)
- Part A: Arm 2 (Placebo+NA [ETV] or [TDF]) (Placebo Comparator): Participants with HBV currently not being treated will receive matching placebo along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: Placebo; Drug: NA (ETV or TDF)
- Part A: Arm 3 (JNJ-56136379 + NA [ETV or TDF]) (Experimental): Participants with HBV currently not being treated will receive JNJ-56136379 along with NA (ETV or TDF) tablet orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: JNJ-56136379; Drug: NA (ETV or TDF)
- Part A: Arm 4 (Placebo + NA [ETV or TDF]) (Placebo Comparator): Virologically suppressed participants will receive matching placebo along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: Placebo; Drug: NA (ETV or TDF)
- Part A: Arm 5 (JNJ-56136379 + NA [ETV or TDF]) (Experimental): Virologically suppressed participants will receive JNJ-56136379 along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: JNJ-56136379; Drug: NA (ETV or TDF)
- Part B: Arm 6 (JNJ-56136379 + NA [ETV or TDF]) (open label) (Experimental): Participants with HBV currently not being treated will receive JNJ-56136379 tablet at a high dose, orally for 24 weeks. The eligible participants may enter the extension phase and will receive JNJ-56136379 along with NA (ETV or TDF) from Week 24 to Week 48.
  Interventions: Drug: JNJ-56136379; Drug: NA (ETV or TDF)
- Part B: Arm 7 (placebo + NA [ETV or TDF]) (Placebo Comparator): Participants with HBV currently not being treated will receive matching placebo along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: Placebo; Drug: NA (ETV or TDF)
- Part B: Arm 8 (JNJ-56136379 + NA [ETV or TDF]) (Experimental): Participants with HBV currently not being treated will receive JNJ-56136379 tablet at a high dose along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: JNJ-56136379; Drug: NA (ETV or TDF)
- Part B: Arm 9 (placebo + NA [ETV or TDF]) (Placebo Comparator): Virologically suppressed participants will receive matching placebo along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: Placebo; Drug: NA (ETV or TDF)
- Part B: Arm 10 (JNJ-56136379 + NA [ETV or TDF]) (Experimental): Virologically suppressed participants will receive JNJ-56136379 tablet at a high dose along with NA (ETV or TDF) tablets orally for 24 weeks. The eligible participants may enter the extension phase and will continue study drugs up to 48 weeks.
  Interventions: Drug: JNJ-56136379; Drug: NA (ETV or TDF)

INTERVENTIONS:
Drug: JNJ-56136379 — Participants will receive JNJ-56136379 tablet orally.
  Other Names: JNJ-6379
  Arms: Part A: Arm 1 (JNJ-56136379 or NA) (open label); Part A: Arm 3 (JNJ-56136379 + NA [ETV or TDF]); Part A: Arm 5 (JNJ-56136379 + NA [ETV or TDF]); Part B: Arm 10 (JNJ-56136379 + NA [ETV or TDF]); Part B: Arm 6 (JNJ-56136379 + NA [ETV or TDF]) (open label); Part B: Arm 8 (JNJ-56136379 + NA [ETV or TDF])
Drug: Placebo — Participants will receive matching placebo tablet orally.
  Arms: Part A: Arm 2 (Placebo+NA [ETV] or [TDF]); Part A: Arm 4 (Placebo + NA [ETV or TDF]); Part B: Arm 7 (placebo + NA [ETV or TDF]); Part B: Arm 9 (placebo + NA [ETV or TDF])
Drug: NA (ETV or TDF) — Participants will receive NA (ETV or TDF) tablet orally as per approved label.

SUMMARY:
The main purpose of this study is to evaluate efficacy of 24 weeks of study treatment, in terms of changes in hepatitis B surface antigen (HBsAg) levels.

DETAILED DESCRIPTION:
The main study consists of 2-parts and each part will consist of 2 types of Chronic Hepatitis B-infected participant populations. Each part of the study will consist of screening phase (up to 8 weeks), treatment phase (24 weeks or 48 weeks, depending on treatment response), and post-treatment follow-up phase (24 weeks or 48 weeks, depending on treatment response). The duration of individual participation will be up to approximately 56 weeks (participants not eligible to continue treatment in extension phase), up to 80 weeks (participants continuing treatment in extension phase but not meeting treatment completion criteria), or up to 104 weeks (participants meeting treatment completion criteria). The safety and efficacy will be monitored throughout the study. In a separate substudy, at selected clinical sites, percutaneous core liver biopsy will be performed to evaluate changes of intrahepatic viral parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (weight in kilogram (kg) divided by the square of height in meters) of 18.0 to 35.0 kilogram / square meter (kg/m^2), extremes included
* Participants must have chronic hepatitis B virus infection (CHB) infection documented by: Serum hepatitis B surface antigen (HBsAg)-positive at screening and serum HBsAg- or hepatitis B virus (HBV) deoxyribonucleic acid (DNA)-positive at least 6 months prior to screening; Serum immunoglobulin M (IgM) anti- hepatitis B core-related (HBc) antibody negative at screening
* In participants currently not being treated (Treatment Arms 1-2-3 and 6-7-8): Participants must not be receiving any CHB treatment at screening, that is, Have never received treatment with HBV antiviral medicines, including NAs or interferon (IFN) products, OR Have not been on treatment with HBV antiviral medicines, including nucleos(t)ide analog (NA)s or IFN products within 6 months prior to baseline (first intake of study drugs), and participants must be HBeAg-positive and have HBV DNA greater than or equal to (>=) 20,000 International Units Per Milliliter (IU/mL), OR be hepatitis B e antigen (HBeAg)-negative and have HBV DNA >=2,000 IU /mL at screening, and participants must have HBsAg greater than (>) 250 IU/mL at screening, and participants must have alanine aminotransferase (ALT) > upper limit of normal (ULN) and less than or equal to (<=) 5 * ULN at screening, determined in the central laboratory
* In virologically suppressed participants (Treatment Arms 4-5 and 9-10): Participants must be virologically suppressed by current NA treatment (entecavir (ETV) or tenofovir disoproxil fumarate (TDF)) as defined by HBV DNA less than (<) 60 IU/mL at screening and at least 6 months prior to screening, and participants must be on the same NA treatment (ETV or TDF) and the same dose for >=12 months prior to screening, and participants must have HBsAg > 250 IU/mL at screening, and participants must have ALT <=2*ULN at screening
* Participants must have: A liver biopsy result classified as Metavir F0-F2 within 1 year prior to screening or at the time of screening, OR FibroScan liver stiffness measurement <8.0 kilopascal (kPa) within 6 months prior to screening or at the time of screening

Exclusion Criteria:

Main Study:

* Participants who test positive for anti-hepatitis B surface (HBs) antibodies
* Participants with current hepatitis A virus infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), hepatitis D virus (HDV) infection (confirmed by HDV antibody), hepatitis E virus infection (confirmed by hepatitis E antibody IgM), or human immunodeficiency virus (HIV)-1 or HIV-2 infection (confirmed by antibodies) at screening; participants with a history of or current HCV infection (confirmed by HCV antibody). Evidence of other active infection (bacterial, viral, fungal, including acute tuberculosis) deemed clinically relevant by the investigator that would interfere with study conduct or its interpretation will also lead to exclusion
* Participants with any evidence of hepatic decompensation at any time point prior to or at the time of screening: Direct bilirubin >1.2* ULN, or International normalized ratio (INR) >1.5* ULN, or Serum albumin < lower limit of normal (LLN), or documented history or current evidence of variceal bleeding, ascites, or hepatic encephalopathy
* Participants with a history of cardiac arrhythmia (example, extrasystoli, tachycardia at rest), history of risk factors for Torsades de Pointes syndrome (example, hypokalemia, family history of long QT syndrome) or history or other clinical evidence of significant or unstable cardiac disease (example, angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, and/or clinically significant 12 lead electrocardiograms (ECGs) abnormalities), moderate to severe valvular disease, or uncontrolled hypertension at screening
* Participants with contraindications to the use of ETV or TDF per local prescribing information

Substudy:

* Presence of coagulopathy or hemoglobinopathy (including sickle cell disease, thalassemia)
* Use of any anti-coagulant, anti-platelet, or non-steroidal anti-inflammatory drug medications from 10 days before until 5 days after each liver biopsy
* Presence of ascites, focal liver lesions, and other findings that would be contraindications for liver biopsies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (76):
- United States (7):
  - The Office of Franco Felizarta, MD, Bakersfield, California
  - Orlando Immunology Center, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Tulane Medical Center (TMC), New Orleans, Louisiana
  - I.D. Care, Inc., Hillsborough, New Jersey
  - NYU Hepatology Associates, New York, New York
  - UPMC Center For Liver Diseases, Pittsburgh, Pennsylvania
- Belgium (3):
  - SGS Clinical Pharmacology Unit (located in ZNA Stuivenberg), Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - GI Research Institute (G.I.R.I.), Vancouver, British Columbia
  - McGill University Health Centre, Montreal, Quebec
  - Toronto General Hospital, Toronto
- China (4):
  - Peking University People's Hospital, Beijing
  - Beiijing Friendship Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Nanfang Hospital, Guangzhou
- France (4):
  - Hôpital Beaujon, Clichy
  - Hopital de La Croix Rousse, Lyon
  - Hopital Saint-Antoine, Paris
  - Hopital Paul Brousse, Villejuif
- Germany (4):
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Johann Wolfgang Goethe- Universität Frankfurt Medizinische Klinik 1, Frankfurt
  - Asklepios Klinik St. Georg, Haus Lifi - Studien und Projekte GmbH, Hamburg
- Hong Kong (2):
  - Queen Mary Hospital, University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, Shatin
- Italy (3):
  - Irccs Ospedale Maggiore Di Milano, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Japan (5):
  - Hiroshima University Hospital, Hiroshima
  - Musashino Red Cross Hospital, Musashino
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - Osaka University Hospital, Suita-shi
- Malaysia (2):
  - Hospital Sultanah Bahiyah, Alor Star
  - University Malaya Medical Centre, Kuala Lumpur
- Poland (4):
  - Szpital Specjalistyczny w Chorzowie, Chorzów
  - Wojewodzki Szpital Zespolony, Kielce
  - ID Clinic, Mysłowice
  - SP ZOZ Wroclawskie Centrum Zdrowia, Wroclaw
- Russia (4):
  - Medical Center SibNovoMed LLC, Novosibirsk
  - Medical Company Hepatolog Ltd, Samara
  - Stavropol State Medical University, Stavropol
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hosp. Clinic I Provincial de Barcelona, Barcelona
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University Hospital, Chiang Mai
  - Prince Of Songkla University, Songkhla
- Turkey (Türkiye) (4):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Saglık Bilimleri University Şişli Trainig and Research Hospital,Department of Gastroenterology, Istanbul
  - Ege University Medical of Faculty, Department of Gastroenterology, Izmir
  - Karadeniz Teknik University Medical Faculty, Trabzon
- Ukraine (4):
  - Kharkiv National Medical University, Regional Clinical Infectious Hospital, Kharkiv
  - SE 'National institute therapy named L.T. Maloi NAMS of Ukraine', Kharkiv
  - Odessa Regional Clinical Hospital, Odesa
  - Vinnytsia City Clinical Hospital #1, Department of Infectious Diseases #1, Vinnytsia
- United Kingdom (4):
  - North Manchester General Hospital, Crumpsall
  - Grahame Hayton Unit, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Verbinnen T, Talloen W, Janssen HLA, Zoulim F, Shukla U, Vandenbossche JJ, Biermer M, De Meyer S, Lenz O. Viral sequence analysis of chronic hepatitis B patients treated with the capsid assembly modulator JNJ-56136379 in the JADE phase 2a study. Antiviral Res. 2023 Aug;216:105660. doi: 10.1016/j.antiviral.2023.105660. Epub 2023 Jun 28. PMID 37385475
- [Derived] Janssen HLA, Hou J, Asselah T, Chan HLY, Zoulim F, Tanaka Y, Janczewska E, Nahass RG, Bourgeois S, Buti M, Lampertico P, Lenz O, Verbinnen T, Vandenbossche J, Talloen W, Kalmeijer R, Beumont M, Biermer M, Shukla U. Randomised phase 2 study (JADE) of the HBV capsid assembly modulator JNJ-56136379 with or without a nucleos(t)ide analogue in patients with chronic hepatitis B infection. Gut. 2023 Jul;72(7):1385-1398. doi: 10.1136/gutjnl-2022-328041. Epub 2023 Jan 25. PMID 36697207
- [Derived] Berke JM, Dehertogh P, Vergauwen K, Mostmans W, Vandyck K, Raboisson P, Pauwels F. Antiviral Properties and Mechanism of Action Studies of the Hepatitis B Virus Capsid Assembly Modulator JNJ-56136379. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02439-19. doi: 10.1128/AAC.02439-19. Print 2020 Apr 21. PMID 32094138

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per planned analysis, the data for Part A Placebo + Nucleos(t)ide analog (NA) and Part B Placebo + NA arm was pooled into a single Placebo + NA arm for data interpretation since there was considerable time overlap in randomization between the two parts, with almost half of the participants of Part B recruited while Part A was still ongoing.
Groups:
- Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] or tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] less than (<) 60 International units per milliliter [IU/mL]) or currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received placebo matching to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg (Open Label): Currently not treated participants received JNJ-56136379 75 mg (3*25 mg tablets) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued treatment with JNJ-56136379 75 mg from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and received treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Virologically suppressed or currently not treated participants received JNJ-56136379 75 mg (3*25 mg tablets) plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg (Open-label): Currently not treated participants received JNJ-56136379 250 mg (2*100 mg and 2*25 mg tablets) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and received treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Virologically suppressed or currently not treated participants received JNJ-56136379 250 mg (2*100 mg and 2*25 mg tablets) plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Period: Overall Study
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open-label) | Part B: JNJ-56136379 250 mg + NA
Started | 43 | 28 | 66 | 32 | 63
Currently Not Treated | 22 | 28 | 33 | 32 | 33
Virologically Suppressed | 21 | 0 | 33 | 0 | 30
Completed | 40 | 24 | 61 | 28 | 58
Not Completed | 3 | 4 | 5 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 0 | 3
Not completed — Disease Relapse | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open-label) | Part B: JNJ-56136379 250 mg + NA | Total
Number analyzed (Participants) | 43 | 28 | 66 | 32 | 63 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (9.53) | 39.2 (12.06) | 40.3 (11.12) | 37.7 (10.92) | 40.5 (10.99) | 40.1 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 20 | 14 | 13 | 70
  Male | 29 | 19 | 46 | 18 | 50 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 42 | 28 | 66 | 32 | 62 | 230
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 11 | 35 | 16 | 30 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 5 | 4 | 1 | 3 | 14
  White | 23 | 11 | 26 | 15 | 30 | 105
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 3 | 2 | 3 | 1 | 2 | 11
  CANADA | 3 | 2 | 3 | 0 | 6 | 14
  CHINA | 1 | 2 | 5 | 4 | 6 | 18
  FRANCE | 3 | 3 | 3 | 0 | 2 | 11
  GERMANY | 3 | 0 | 0 | 2 | 4 | 9
  ITALY | 4 | 1 | 3 | 1 | 1 | 10
  JAPAN | 1 | 0 | 2 | 2 | 3 | 8
  MALAYSIA | 1 | 2 | 1 | 1 | 3 | 8
  POLAND | 4 | 1 | 7 | 0 | 6 | 18
  RUSSIAN FEDERATION | 4 | 1 | 4 | 3 | 6 | 18
  SOUTH KOREA | 1 | 1 | 2 | 1 | 2 | 7
  SPAIN | 2 | 1 | 6 | 1 | 2 | 12
  TAIWAN | 5 | 4 | 18 | 1 | 4 | 32
  THAILAND | 1 | 0 | 0 | 3 | 3 | 7
  TURKEY | 2 | 6 | 6 | 4 | 5 | 23
  UKRAINE | 1 | 0 | 0 | 5 | 4 | 10
  UNITED KINGDOM | 2 | 2 | 2 | 2 | 2 | 10
  UNITED STATES | 2 | 0 | 1 | 0 | 2 | 5
  Hong Kong | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatitis B Surface Antigen (HBsAg) Levels in Currently Not Treated Population at Week 24
Description: Change from baseline in HBsAg levels in currently not treated population at Week 24 based on Hepatitis B e Antigen (HBeAg) status was reported. Currently not treated population defined as participants who didn't receive any hepatitis B virus (HBV) treatment 6 months prior to baseline.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat Population (ITT) consisted of all participants who were randomized and received at least one dose of any study agent. If a participant received a study agent other than their randomly assigned study agent, participants were shown in the treatment arm as randomized. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n'(number analyzed) represents number of participants evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: log10 IU per milliliter (log10 IU/mL)
Groups:
- Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg (Open Label): Currently not treated participants received 3*25 mg tablets of JNJ-56136379 once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued treatment with JNJ-56136379 75 mg from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and received treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg (Open Label): Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and received treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 21 | 33 | 30 | 30
log10 IU per milliliter (log10 IU/mL)
  HBeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  HBeAg Positive | -0.251 (0.3144) | -0.096 (0.3567) | -0.142 (0.3443) | -0.203 (0.4721) | -0.411 (0.4843)
  HBeAg Negative: number analyzed (Participants) | 13 | 13 | 21 | 16 | 19
  HBeAg Negative | 0.015 (0.0880) | 0.053 (0.2066) | 0.041 (0.0939) | 0.064 (0.0913) | 0.088 (0.1613)

2. Primary Outcome: Change From Baseline in HBsAg Levels in Virologically Suppressed Population at Week 24
Description: Change from baseline in HBsAg levels in virologically suppressed population at Week 24 based on HBeAg status was reported. Virologically suppressed population defined as participants who were on entecavir (ETV) or tenofovir disoproxil fumarate (TDF) for at least 12 months prior to screening and had HBV deoxyribonucleic acid (DNA) <60 IU/mL. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Baseline and Week 24
Population: ITT population consisted of all participants who were randomized and received at least one dose of any study agent. If a participant received a study agent other than their randomly assigned study agent, participants were shown in the treatment arm as randomized. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] or tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) participants received matching placebo to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Virologically suppressed participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Virologically suppressed participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 29
log10 IU/mL
  HBeAg Positive: number analyzed (Participants) | 5 | 9 | 10
  HBeAg Positive | 0.008 (0.1224) | -0.063 (0.2272) | 0.105 (0.1809)
  HBeAg Negative: number analyzed (Participants) | 15 | 24 | 19
  HBeAg Negative | 0.024 (0.0722) | -0.017 (0.0677) | 0.092 (0.0556)

3. Secondary Outcome: Number of Participants With Treatment- Emergent Adverse Events (AEs)
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Treatment-emergent AEs were AEs with onset during the treatment phase or that worsened since baseline.
Time Frame: Up to Week 48
Population: The safety population included all participants who received at least one dose of the study agent; all safety endpoints were analyzed by the treatment arm as treated.
Measure: Count of Participants; unit: Participants
Groups:
- Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] or tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) or currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Virologically suppressed or currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Virologically suppressed or currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 43 | 28 | 66 | 32 | 63
Participants | 34 | 18 | 55 | 25 | 54

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Week 80
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 43 | 28 | 66 | 32 | 63
Participants | 1 | 1 | 4 | 0 | 4

5. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs, Physical Examinations, Electrocardiogram (ECG), and Clinical Laboratory Tests
Description: Number of participants with clinically significant changes in vital signs, physical examinations, ECG, and clinical laboratory tests (including hematology, blood biochemistry, blood coagulation, and urinalysis) were reported.
Time Frame: Up to Week 80
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 43 | 28 | 66 | 32 | 63
Participants
  Vital Signs | 0 | 0 | 0 | 0 | 0
  Physical Examinations | 0 | 0 | 0 | 0 | 0
  ECG | 0 | 0 | 0 | 0 | 0
  Clinical Laboratory Tests: Hematology | 0 | 0 | 0 | 0 | 0
  Clinical Laboratory Tests: Blood biochemistry | 0 | 0 | 0 | 0 | 0
  Clinical Laboratory Tests: Blood coagulation | 0 | 0 | 0 | 0 | 0
  Clinical Laboratory Tests: Urinalysis | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in HBsAg Levels in Currently Not Treated Population Over Time
Description: Change from baseline in HBsAg levels in currently not treated population based on HBeAg status was reported.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 23 | 33 | 30 | 30
log10 IU/mL
  Week 24: HBeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: HBeAg Positive | -0.251 (0.3144) | -0.096 (0.3567) | -0.142 (0.3443) | -0.203 (0.4721) | -0.411 (0.4843)
  Week 24: HBeAg Negative: number analyzed (Participants) | 13 | 13 | 21 | 16 | 19
  Week 24: HBeAg Negative | 0.015 (0.0880) | 0.053 (0.2066) | 0.041 (0.0939) | 0.064 (0.0913) | 0.088 (0.1613)
  Week 48: HBeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HBeAg Positive | -0.109 (0.2065) |  | 0.061 (0.6817) | -0.035 (0.6065) | -0.811 (1.0053)
  Week 48: HBeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HBeAg Negative | 0.027 (0.0969) |  | -0.024 (0.1016) | 0.011 (0.1086) | 0.075 (0.1528)
  Follow-up Week 24: HBeAg Positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: HBeAg Positive | -0.300 (0.3333) | -0.786 (0.6879) | -0.404 (0.5852) | -0.230 (0.5110) | -0.721 (0.5666)
  Follow-up Week 24: HBeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24: HBeAg Negative | 0.006 (0.1191) | 0.000 (0.1889) | -0.068 (0.0999) | -0.073 (0.1195) | -0.017 (0.1533)

7. Secondary Outcome: Change From Baseline in HBsAg Levels in Virologically Suppressed Population Over Time
Description: Change from baseline in HBsAg levels in virologically suppressed population based on HBeAg status was reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 29
log10 IU/mL
  Week 24: HBeAg Positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: HBeAg Positive | 0.008 (0.1224) | -0.063 (0.2272) | 0.105 (0.1809)
  Week 24: HBeAg Negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HBeAg Negative | 0.024 (0.0722) | -0.017 (0.0677) | 0.092 (0.0556)
  Week 48: HBeAg Positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: HBeAg Positive | 0.043 (0.1374) | -0.078 (0.2660) | 0.046 (0.2223)
  Week 48: HBeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: HBeAg Negative | 0.011 (0.0736) | -0.038 (0.0747) | 0.029 (0.0752)
  Follow-up Week 24: HBeAg Positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: HBeAg Positive | -0.088 (0.0492) | -0.146 (0.2821) | -0.159 (0.2141)
  Follow-up Week 24: HBeAg Negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: HBeAg Negative | -0.006 (0.0789) | -0.119 (0.1172) | -0.028 (0.0655)

8. Secondary Outcome: Percentage of Participants With HBsAg Levels Less Than (<) 1,000 or <100 International Units Per Milliliter (IU/mL) in Currently Not Treated Population
Description: Percentage of participants with HBsAg levels <1,000 or <100 IU/mL in currently not treated population based on their HBeAg status were reported.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 23 | 33 | 30 | 30
Percentage of participants
  Week 24: HBsAg<100 IU/mL: HBeAg positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: HBsAg<100 IU/mL: HBeAg positive | 0 | 0 | 0 | 0 | 0
  Week 24: HBsAg<1000 IU/mL: HBeAg positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: HBsAg<1000 IU/mL: HBeAg positive | 0 | 0 | 8.3 | 0 | 0
  Week 24: HBsAg<100 IU/mL: HBeAg negative: number analyzed (Participants) | 13 | 13 | 21 | 16 | 19
  Week 24: HBsAg<100 IU/mL: HBeAg negative | 0 | 0 | 0 | 0 | 0
  Week 24: HBsAg<1000 IU/mL: HBeAg negative: number analyzed (Participants) | 13 | 13 | 21 | 16 | 19
  Week 24: HBsAg<1000 IU/mL: HBeAg negative | 15.4 | 23.1 | 4.8 | 0 | 10.5
  Week 48: HBsAg<100 IU/mL: HBeAg positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HBsAg<100 IU/mL: HBeAg positive | 0 |  | 0 | 0 | 0
  Week 48: HBsAg<1000 IU/mL: HBeAg positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HBsAg<1000 IU/mL: HBeAg positive | 0 |  | 50.0 | 0 | 20.0
  Week 48: HBsAg<100 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HBsAg<100 IU/mL: HBeAg Negative | 0 |  | 0 | 0 | 0
  Week 48: HBsAg<1000 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HBsAg<1000 IU/mL: HBeAg Negative | 18.2 |  | 22.2 | 7.7 | 14.3
  Follow-up Week 24:HBsAg<100 IU/mL: HBeAg Positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24:HBsAg<100 IU/mL: HBeAg Positive | 0 | 0 | 0 | 0 | 0
  Follow-up Week 24:HBsAg<1000 IU/mL: HBeAg positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24:HBsAg<1000 IU/mL: HBeAg positive | 0 | 10.0 | 8.3 | 0 | 9.1
  Follow-up Week 24:HBsAg<100 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24:HBsAg<100 IU/mL: HBeAg Negative | 0 | 0 | 0 | 0 | 0
  Follow-up Week 24: HBsAg<1000 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24: HBsAg<1000 IU/mL: HBeAg Negative | 18.2 | 23.1 | 18.8 | 7.1 | 5.9

9. Secondary Outcome: Percentage of Participants With HBsAg Levels <1,000 or <100 IU/mL in Virologically Suppressed Population
Description: Percentage of participants with HBsAg levels <1,000 or <100 IU/mL in virologically suppressed population based on their HBeAg status were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 29
Percentage of participants
  Week 24: HBsAg<100 IU/mL: HBeAg positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: HBsAg<100 IU/mL: HBeAg positive | 0 | 0 | 0
  Week 24: HBsAg<1000 IU/mL: HBeAg positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: HBsAg<1000 IU/mL: HBeAg positive | 20.0 | 11.1 | 10.0
  Week 24: HBsAg<100 IU/mL: HBeAg negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HBsAg<100 IU/mL: HBeAg negative | 0 | 0 | 0
  Week 24: HBsAg<1000 IU/mL: HBeAg negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HBsAg<1000 IU/mL: HBeAg negative | 0 | 29.2 | 15.8
  Week 48: HBsAg<100 IU/mL: HBeAg positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: HBsAg<100 IU/mL: HBeAg positive | 0 | 0 | 0
  Week 48: HBsAg<1000 IU/mL: HBeAg positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: HBsAg<1000 IU/mL: HBeAg positive | 20.0 | 12.5 | 33.3
  Week 48: HBsAg<100 IU/mL: HBeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: HBsAg<100 IU/mL: HBeAg Negative | 0 | 0 | 0
  Week 48: HBsAg<1000 IU/mL: HBeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: HBsAg<1000 IU/mL: HBeAg Negative | 7.7 | 33.3 | 20.0
  Follow-up Week 24: HBsAg<100 IU/mL: HBeAg positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: HBsAg<100 IU/mL: HBeAg positive | 0 | 11.1 | 0
  Follow-up Week 24: HBsAg<1000 IU/mL: HBeAg positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: HBsAg<1000 IU/mL: HBeAg positive | 25.0 | 11.1 | 44.4
  Follow-up Week 24: HBsAg<100 IU/mL: HBeAg negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: HBsAg<100 IU/mL: HBeAg negative | 0 | 0 | 0
  Follow-up Week 24: HBsAg<1000 IU/mL: HBeAg negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: HBsAg<1000 IU/mL: HBeAg negative | 13.3 | 34.8 | 7.1

10. Secondary Outcome: Percentage of Participants With Greater Than (>) 0.5 log10 IU/mL or >1 log10 IU/mL Reduction in HBsAg From Baseline in Currently Not Treated Population
Description: Percentage of participants with >0.5 log10 IU/mL or >1 log10 IU/mL reduction in HBsAg from baseline in currently not treated population based on their HBeAg status were reported.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 23 | 33 | 30 | 30
Percentage of participants
  Week 24: >0.5 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: >0.5 log10 IU/mL: HBeAg Positive | 12.5 | 12.5 | 8.3 | 28.6 | 36.4
  Week 24: >1 log10IU/mL: HBeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: >1 log10IU/mL: HBeAg Positive | 0 | 0 | 0 | 7.1 | 18.2
  Week 24: >0.5 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 13 | 13 | 21 | 16 | 19
  Week 24: >0.5 log10 IU/mL: HBeAg Negative | 0 | 0 | 0 | 0 | 0
  Week 24: >1 log10 IU/mL: Negative: number analyzed (Participants) | 13 | 13 | 21 | 16 | 19
  Week 24: >1 log10 IU/mL: Negative | 0 | 0 | 0 | 0 | 0
  Week 48: >0.5 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: >0.5 log10 IU/mL: HBeAg Positive | 0 |  | 0 | 20.0 | 60.0
  Week 48: >1 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: >1 log10 IU/mL: HBeAg Positive | 0 |  | 0 | 0 | 60.0
  Week 48: >0.5 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: >0.5 log10 IU/mL: HBeAg Negative | 0 |  | 0 | 0 | 0
  Week 48: >1 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: >1 log10 IU/mL: HBeAg Negative | 0 |  | 0 | 0 | 0
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Positive | 14.3 | 60.0 | 33.3 | 30.0 | 54.5
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Positive | 0 | 40.0 | 16.7 | 7.7 | 27.3
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Negative | 0 | 0 | 0 | 0 | 0
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Negative | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With >0.5 log10 IU/mL or >1 log10 IU/mL Reduction in HBsAg From Baseline in Virologically Suppressed Population
Description: Percentage of participants with >0.5 log10 IU/mL or >1 log10 IU/mL reduction in HBsAg from baseline in virologically suppressed population based on their HBeAg status were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 29
Percentage of participants
  Week 24: >0.5 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: >0.5 log10 IU/mL: HBeAg Positive | 0 | 0 | 0
  Week 24: >1 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: >1 log10 IU/mL: HBeAg Positive | 0 | 0 | 0
  Week 24: >0.5 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: >0.5 log10 IU/mL: HBeAg Negative | 0 | 0 | 0
  Week 24: >1 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: >1 log10 IU/mL: HBeAg Negative | 0 | 0 | 0
  Week 48: >0.5 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: >0.5 log10 IU/mL: HBeAg Positive | 0 | 12.5 | 0
  Week 48: >1 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: >1 log10 IU/mL: HBeAg Positive | 0 | 0 | 0
  Week 48: >0.5 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: >0.5 log10 IU/mL: HBeAg Negative | 0 | 0 | 0
  Week 48: >1 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: >1 log10 IU/mL: HBeAg Negative | 0 | 0 | 0
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Positive | 0 | 11.1 | 11.1
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Positive | 0 | 0 | 0
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: >0.5 log10 IU/mL: HBeAg Negative | 0 | 0 | 0
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: >1 log10 IU/mL: HBeAg Negative | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels in Currently Not Treated Population
Description: Change from baseline in HBV DNA levels in currently not treated population based on their HBeAg status was reported.
Time Frame: Baseline up to Weeks 24, 48 and Follow-up Week 24
Population: ITT population consisted of all participants who are randomized and received at least one dose of any study agent. If a participant received a study agent other than their randomly assigned study agent, participants would be shown in the treatment arm as randomized. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 22 | 33 | 30 | 30
log10 IU/mL
  Week 24: HbeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: HbeAg Positive | -5.211 (1.1986) | -3.284 (2.1148) | -5.531 (0.7915) | -5.719 (0.8395) | -5.883 (1.1396)
  Week 24:HbeAg Negative: number analyzed (Participants) | 13 | 14 | 21 | 16 | 19
  Week 24:HbeAg Negative | -3.622 (1.3003) | -3.469 (1.2901) | -4.077 (0.9435) | -3.545 (1.1482) | -3.690 (1.5289)
  Week 48: HbeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HbeAg Positive | -6.359 (0.1989) |  | -5.009 (1.8289) | -6.413 (0.9121) | -6.205 (1.3358)
  Week 48: HbeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HbeAg Negative | -3.650 (1.3342) |  | -3.707 (1.6444) | -3.313 (1.0138) | -3.520 (1.2505)
  Follow-up Week 24: HbeAg Positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: HbeAg Positive | -5.956 (0.6580) | -6.318 (1.0238) | -6.080 (0.8678) | -6.262 (0.6278) | -6.013 (1.8359)
  Follow-up Week 24: HbeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24: HbeAg Negative | -3.727 (1.6598) | -4.805 (1.0557) | -4.165 (1.1102) | -3.721 (1.1937) | -3.906 (1.6486)

13. Secondary Outcome: Change From Baseline in HBV DNA Levels in Virologically Suppressed Population
Description: Change from baseline in HBV DNA levels in virologically supressed population based on their HBeAg status was reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Baseline up to Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 29
log10 IU/mL
  Week 24: HbeAg Positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: HbeAg Positive | -0.051 (0.1142) | 0.000 (0.3374) | 0.021 (0.2665)
  Week 24: HbeAg Negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HbeAg Negative | -0.032 (0.2184) | 0.016 (0.3626) | -0.024 (0.2472)
  Week 48: HbeAg Positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: HbeAg Positive | 0.044 (0.2660) | 0.000 (0.3607) | -0.233 (0.2817)
  Week 48: HbeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: HbeAg Negative | 0.000 (0.3896) | -0.010 (0.3403) | -0.093 (0.2645)
  Follow-up Week 24: HbeAg Positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: HbeAg Positive | 0.175 (0.3644) | 0.000 (0.3374) | 0.105 (0.5370)
  Follow-up Week 24: HbeAg Negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: HbeAg Negative | -0.032 (0.2832) | -0.069 (0.3767) | 0.070 (0.3124)

14. Secondary Outcome: Percentage of Participants With Undetectable HBV DNA Levels in Currently Not Treated Population
Description: Percentage of participants with undetectable HBV DNA levels in currently not treated population based on their HBeAg status was evaluated.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: ITT population consisted of all participants who were randomized and received at least one dose of any study agent. If a participant received a study agent other than their randomly assigned study agent, participants were shown in the treatment arm as randomized. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure 'n' (number analyzed) represents number of participants evaluable for the specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 23 | 33 | 30 | 30
Percentage of participants
  Week 24: HBeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: HBeAg Positive | 0 | 0 | 0 | 0 | 9.1
  Week 24: HBeAg Negative: number analyzed (Participants) | 13 | 14 | 21 | 16 | 19
  Week 24: HBeAg Negative | 23.1 | 14.3 | 14.3 | 18.8 | 0
  Week 48: HBeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HBeAg Positive | 0 |  | 20.0 | 0 | 0
  Week 48: HBeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HBeAg Negative | 27.3 |  | 55.6 | 15.4 | 28.6
  Follow-up Week 24: HBeAg Positive: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: HBeAg Positive | 0 | 0 | 0 | 15.4 | 11.9
  Follow-up Week 24: HBeAg Negative: number analyzed (Participants) | 11 | 13 | 16 | 14 | 17
  Follow-up Week 24: HBeAg Negative | 36.4 | 38.5 | 18.8 | 35.7 | 23.5

15. Secondary Outcome: Percentage of Participants With Undetectable HBV DNA Levels in Virologically Suppressed Population
Description: Percentage of participants with undetectable HBV DNA levels in virologically suppressed population based on their HBeAg status were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] or tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml)) participants received matching placebo to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 29
Percentage of participants
  Week 24: HBeAg positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: HBeAg positive | 40.0 | 22.2 | 40.0
  Week 24: HBeAg negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HBeAg negative | 60.0 | 58.3 | 63.2
  Week 48: HBeAg positive: number analyzed (Participants) | 5 | 8 | 9
  Week 48: HBeAg positive | 40.0 | 37.5 | 77.8
  Week 48: HBeAg negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: HBeAg negative | 53.8 | 66.7 | 66.7
  Follow-up Week 24: HBeAg positive: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: HBeAg positive | 25.0 | 44.4 | 44.4
  Follow-up Week 24: HBeAg negative: number analyzed (Participants) | 15 | 23 | 14
  Follow-up Week 24: HBeAg negative | 60.0 | 73.9 | 42.9

16. Secondary Outcome: Change From Baseline in HBeAg Levels in Currently Not Treated Population
Description: Change from baseline in HBeAg levels in HBeAg positive currently not treated population was reported.
Time Frame: Baseline up to Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 8 | 10 | 12 | 14 | 11
log10 IU/mL
  Week 24: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24 | -0.811 (0.7953) | -0.456 (0.2908) | -0.487 (2974) | -0.974 (0.8400) | -0.701 (0.6645)
  Week 48: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48 | -2.250 (0.4010) |  | -0.235 (0.0908) | -1.779 (1.3525) | -1.601 (1.2689)
  Follow-up Week 24: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24 | -1.139 (1.2528) | -1.597 (1.1587) | -0.876 (0.5178) | -1.243 (0.9933) | -1.215 (1.2910)

17. Secondary Outcome: Change From Baseline in HBeAg Levels in Virologically Suppressed Population
Description: Change from baseline in HBeAg levels in HBeAg positive virologically suppressed population was reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Baseline up to Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Part A: JNJ-56136379 75 mg + NA: Virologically suppressed received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 5 | 9 | 10
log10 IU/mL
  Week 24 | -0.313 (0.5281) | -0.315 (0.4681) | -0.162 (0.2037)
  Week 48: number analyzed (Participants) | 5 | 8 | 9
  Week 48 | -0.589 (0.6616) | -0.393 (0.4866) | -0.291 (0.2376)
  Follow-up Week 24: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24 | -0.772 (0.7059) | -0.387 (0.5218) | -0.351 (0.2877)

18. Secondary Outcome: Percentage of Participants With >0.5 log10 IU/mL and >1 log10 IU/mL Reduction in HBeAg From Baseline in Currently Not Treated Population
Description: Percentage of participants with >0.5 log10 IU/mL and >1 log10 IU/mL reduction in HBeAg from baseline in HBeAg positive currently not treated population was reported.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 8 | 10 | 12 | 14 | 11
Percentage of participants
  Week 24: >0.5 log10 IU/mL: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: >0.5 log10 IU/mL | 62.5 | 50 | 41.7 | 78.6 | 63.6
  Week 24: >1 log10 IU/mL: number analyzed (Participants) | 8 | 8 | 12 | 14 | 11
  Week 24: >1 log10 IU/mL | 37.5 | 0 | 8.3 | 42.9 | 36.4
  Week 48: >0.5 log10 IU/mL: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: >0.5 log10 IU/mL | 100 |  | 0 | 100.0 | 80.0
  Week 48: >1 log10 IU/mL: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: >1 log10 IU/mL | 100.0 |  | 0 | 80.0 | 80.0
  Follow-up Week 24: >0.5 log10 IU/mL: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: >0.5 log10 IU/mL | 42.9 | 80.0 | 91.7 | 84.6 | 72.7
  Follow-up Week 24: >1 log10 IU/mL: number analyzed (Participants) | 7 | 10 | 12 | 13 | 11
  Follow-up Week 24: >1 log10 IU/mL | 28.6 | 70.0 | 25.0 | 61.5 | 45.5

19. Secondary Outcome: Percentage of Participants With >0.5 log10 IU/mL and >1 log10 IU/mL Reduction in HBeAg From Baseline in Virologically Suppressed Population
Description: Percentage of participants with >0.5 log10 IU/mL and >1 log10 IU/mL reduction in HBeAg from baseline in HBeAg positive virologically suppressed population was reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 5 | 9 | 10
Percentage of participants
  Week 24: >0.5 log10 IU/mL | 20 | 33.3 | 10
  Week 24: >1 log10 IU/mL | 20 | 11.1 | 0
  Week 48: >0.5 log10 IU/mL: number analyzed (Participants) | 5 | 8 | 9
  Week 48: >0.5 log10 IU/mL | 20.0 | 25.0 | 22.2
  Week 48: >1 log10 IU/mL: number analyzed (Participants) | 5 | 8 | 9
  Week 48: >1 log10 IU/mL | 20.0 | 25.0 | 0
  Follow-up Week 24: >0.5 log10 IU/mL: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: >0.5 log10 IU/mL | 50.0 | 22.2 | 22.2
  Follow-up Week 24: >1 log10 IU/mL: number analyzed (Participants) | 4 | 9 | 9
  Follow-up Week 24: >1 log10 IU/mL | 25.0 | 11.1 | 0

20. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance in Currently Not Treated Population
Description: Percentage of participants with HBsAg seroclearance in currently not treated population based on their HBeAg status were reported. Seroclearance at Week 24/48 of the treatment defined as a confirmed loss of HBsAg at Week 24/48. Loss is defined as a baseline HBsAg with a repeat reactive, confirmed or positive result and a post-baseline assessment with a negative result. This outcome measure was planned to be analyzed at specified timepoints only.
Time Frame: Weeks 24 and 48
Population: ITT population consisted of all participants who were randomized and received at least one dose of any study agent. If a participant received a study agent other than their randomly assigned study agent, participants were shown in the treatment arm as randomized. Here, 'n' (number analyzed) represents number of participants evaluable for the specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 20 | 33 | 29 | 28
Percentage of participants
  Week 24: HbeAg Positive: number analyzed (Participants) | 8 | 8 | 12 | 14 | 10
  Week 24: HbeAg Positive | 0 | 0 | 0 | 0 | 0
  Week 24: HbeAg Negative: number analyzed (Participants) | 13 | 12 | 21 | 15 | 18
  Week 24: HbeAg Negative | 0 | 0 | 0 | 0 | 0
  Week 48: HbeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HbeAg Positive | 0 |  | 0 | 20.0 | 0
  Week 48: HbeAg Negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HbeAg Negative | 0 |  | 0 | 0 | 0

21. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance in Virologically Suppressed Population
Description: Percentage of participants with HBsAg seroclearance in virologically suppressed population based on their HBeAg status were reported. Seroclearance at Week 24/48 of the treatment defined as a confirmed loss of HBsAg at Week 24/48. Loss is defined as a baseline HBsAg with a repeat reactive, confirmed or positive result and a post-baseline assessment with a negative result. This outcome measure was planned to be analyzed for specified arms and specific timepoints only .
Time Frame: Weeks 24 and 48
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 20 | 33 | 30
Percentage of participants
  Week 24: HbeAg Positive: number analyzed (Participants) | 5 | 9 | 10
  Week 24: HbeAg Positive | 0 | 0 | 0
  Week 24: HbeAg Negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HbeAg Negative | 0 | 0 | 0
  Week 48: HbeAg Positive: number analyzed (Participants) | 5 | 9 | 9
  Week 48: HbeAg Positive | 20.0 | 0 | 0
  Week 48: HbeAg Negative: number analyzed (Participants) | 13 | 21 | 15
  Week 48: HbeAg Negative | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion in Currently Not Treated Population
Description: Percentage of participants with HBsAg seroconversion in currently not treated population based on their HBeAg status were reported. Seroconversion at Week 24/48 of the treatment defined as a confirmed loss of HBsAg at week 24/48 of the treatment and an appearance of Anti-HBs. This outcome measure was planned to be analyzed for specified timepoints only.
Time Frame: Weeks 24 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Part B: JNJ-56136379 250 mg + NA: Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase.Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 20 | 32 | 28 | 28
Percentage of participants
  Week 24: HbeAg Positive: number analyzed (Participants) | 8 | 8 | 11 | 13 | 10
  Week 24: HbeAg Positive | 0 | 0 | 0 | 0 | 0
  Week 24: HbeAg negative: number analyzed (Participants) | 13 | 12 | 21 | 15 | 18
  Week 24: HbeAg negative | 0 | 0 | 0 | 0 | 0
  Week 48: HbeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HbeAg Positive | 0 |  | 0 | 0 | 0
  Week 48: HbeAg negative: number analyzed (Participants) | 11 | 0 | 9 | 13 | 14
  Week 48: HbeAg negative | 0 |  | 0 | 0 | 0

23. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion in Virologically Suppressed Population
Description: Percentage of participants with HBsAg seroconversion in virologically suppressed population based on their HBeAg status were reported. Seroconversion at Week 24/48 of the treatment defined as a confirmed loss of HBsAg at week 24/48 of the treatment and an appearance of Anti-HBs. This outcome measure was planned to be analyzed for specified arms and specified timepoints only.
Time Frame: Weeks 24 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 33 | 29
Percentage of participants
  Week 24: HbeAg Positive: number analyzed (Participants) | 6 | 9 | 10
  Week 24: HbeAg Positive | 0.0 | 0.0 | 0.0
  Week 24: HbeAg negative: number analyzed (Participants) | 15 | 24 | 19
  Week 24: HbeAg negative | 0.0 | 0.0 | 0.0
  Week 48: HbeAg Positive: number analyzed (Participants) | 9 | 5 | 8
  Week 48: HbeAg Positive | 0.0 | 0.0 | 0.0
  Week 48: HbeAg negative: number analyzed (Participants) | 10 | 21 | 15
  Week 48: HbeAg negative | 0.0 | 0.0 | 0.0

24. Secondary Outcome: Percentage of Participants With Normalized Alanine Aminotransferase (ALT) Levels in Currently Not Treated Population
Description: Percentage of participants with normalized ALT levels in currently not treated population, whose ALT levels were above upper limit of normal at baseline based on their HBeAg status were reported.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: The safety population included all participants who received at least one dose of the study agent with ALT values higher than upper limit of normal (ULN) at baseline if time point is available; all safety endpoints were analyzed by the treatment arm as treated. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable for the specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 17 | 19 | 27 | 25 | 24
Percentage of participants
  Week 24: HBeAg positive: number analyzed (Participants) | 8 | 5 | 11 | 14 | 9
  Week 24: HBeAg positive | 62.5 | 60.0 | 54.5 | 64.3 | 44.4
  Week 24: HBeAg negative: number analyzed (Participants) | 9 | 12 | 16 | 11 | 15
  Week 24: HBeAg negative | 55.6 | 91.7 | 68.8 | 72.7 | 80.0
  Week 48: HBeAg positive: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5
  Week 48: HBeAg positive | 100.0 |  | 100.0 | 60.0 | 40.0
  Week 48: HBeAg negative: number analyzed (Participants) | 8 | 0 | 6 | 9 | 11
  Week 48: HBeAg negative | 75.0 |  | 100.0 | 77.8 | 63.6
  Follow-up Week 24: HBeAg positive: number analyzed (Participants) | 7 | 7 | 11 | 13 | 9
  Follow-up Week 24: HBeAg positive | 71.4 | 71.4 | 63.6 | 61.5 | 77.8
  Follow-up Week 24: HBeAg negative: number analyzed (Participants) | 8 | 12 | 12 | 11 | 15
  Follow-up Week 24: HBeAg negative | 87.5 | 100.0 | 83.3 | 90.9 | 86.7

25. Secondary Outcome: Percentage of Participants With Normalized ALT Levels in Virologically Suppressed Population
Description: Percentage of participants with normalized ALT levels in virologically suppressed population, whose ALT levels were above upper limit of normal at baseline based on their HBeAg status were reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24, 48 and Follow-up Week 24
Population: The safety population included all participants who received at least one dose of the study agent with ALT values higher than ULN at baseline if time point is available; all safety endpoints were analyzed by the treatment arm as treated. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable for the specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 2 | 4 | 5
Percentage of participants
  Week 24: HBeAg Positive: number analyzed (Participants) | 0 | 1 | 3
  Week 24: HBeAg Positive |  | 100.0 | 33.3
  Week 24: HBeAg Negative: number analyzed (Participants) | 2 | 3 | 2
  Week 24: HBeAg Negative | 50.0 | 100.0 | 0
  Week 48: HBeAg positive: number analyzed (Participants) | 0 | 1 | 3
  Week 48: HBeAg positive |  | 100.0 | 33.3
  Week 48: HBeAg negative: number analyzed (Participants) | 2 | 2 | 2
  Week 48: HBeAg negative | 50.0 | 0 | 50.0
  Follow-up Week 24: HBeAg Positive: number analyzed (Participants) | 0 | 1 | 3
  Follow-up Week 24: HBeAg Positive |  | 100.0 | 33.3
  Follow-up Week 24: HBeAg negative: number analyzed (Participants) | 2 | 3 | 1
  Follow-up Week 24: HBeAg negative | 50.0 | 66.7 | 100.0

26. Secondary Outcome: Percentage of Participants With Virological Breakthrough in Currently Not Treated Population
Description: Percentage of participants with virological breakthrough in currently not treated population based on their HBeAg status was reported. Virological breakthrough defined as confirmed on treatment HBV DNA increase by >1 log10 from nadir level or confirmed on treatment level >200 IU/mL in participants who had HBV DNA level below the lower limit of quantification (LLOQ) of the HBV DNA assay.
Time Frame: Weeks 24 and 48
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 22 | 28 | 33 | 32 | 33
Percentage of participants
  Week 24: HbeAg Positive: number analyzed (Participants) | 8 | 12 | 12 | 14 | 13
  Week 24: HbeAg Positive | 0 | 16.7 | 0 | 0 | 0
  Week 24: HbeAg Negative: number analyzed (Participants) | 14 | 16 | 21 | 18 | 20
  Week 24: HbeAg Negative | 0 | 18.8 | 0 | 5.6 | 0
  Week 48: HbeAg Positive: number analyzed (Participants) | 2 | 0 | 2 | 6 | 5
  Week 48: HbeAg Positive | 100.0 |  | 100.0 | 100.0 | 100.0
  Week 48: HbeAg Negative: number analyzed (Participants) | 12 | 3 | 10 | 14 | 16
  Week 48: HbeAg Negative | 0 | 33.3 | 10.0 | 0 | 0

27. Secondary Outcome: Percentage of Participants With Virological Breakthrough in Virologically Suppressed Population
Description: Percentage of participants with virological breakthrough in virologically suppressed population based on their HBeAg status was reported. Virological breakthrough defined as confirmed on treatment HBV DNA increase by >1 log10 from nadir level or confirmed on treatment level >200 IU/mL in participants who had HBV DNA level below the lower limit of quantification (LLOQ) of the HBV DNA assay. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Weeks 24 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 21 | 33 | 30
Percentage of participants
  Week 24: HbeAg Positive: number analyzed (Participants) | 6 | 9 | 10
  Week 24: HbeAg Positive | 0 | 0 | 0
  Week 24: HbeAg Negative: number analyzed (Participants) | 15 | 24 | 20
  Week 24: HbeAg Negative | 0 | 0 | 0
  Week 48: HbeAg Positive: number analyzed (Participants) | 5 | 8 | 10
  Week 48: HbeAg Positive | 0 | 0 | 0
  Week 48: HbeAg Negative: number analyzed (Participants) | 14 | 23 | 17
  Week 48: HbeAg Negative | 0 | 0 | 0

28. Secondary Outcome: Plasma Concentrations of Entecavir [ETV] in Currently Not Treated Population
Description: Plasma concentrations of ETV administered as monotherapy or co-administered with JNJ-56136379 in currently not treated population was determined. As planned, plasma concentration of ETV co-administered with placebo was analyzed separately for Part A and Part B. Samples were analyzed using POP PK modeling.
Time Frame: Day 1: 0 hours, 2 hours; Weeks 1, 2, 4, 8, 12, 20, 24, 28, 32, 36, 44, 48: 0 hours; Follow-up: Weeks 2 and 4
Population: The pharmacokinetic (PK) analysis set included data for all participants with available plasma concentrations. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA): Currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (75 milligrams [mg]) plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part B: Placebo (Matching to JNJ-56136379 250 mg) + Nucleos(t)Ide Analog (NA): Currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (250 mg) plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
Arm/Group | Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA) | Part B: Placebo (Matching to JNJ-56136379 250 mg) + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 1 | 3 | 6 | 7
nanograms per milliliter (ng/mL)
  Day 1: 0 hours: number analyzed (Participants) | 0 | 0 | 2 | 4
  Day 1: 0 hours |  |  | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point.
  Day 1: 2 hours: number analyzed (Participants) | 1 | 2 | 4 | 3
  Day 1: 2 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 1.39 (0.709) | 1.18 (0.197)
  Week 1: 0 hours: number analyzed (Participants) | 1 | 3 | 5 | 6
  Week 1: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.321 (0.0961) | 0.289 (0.0351)
  Week 2: 0 hours: number analyzed (Participants) | 1 | 2 | 5 | 7
  Week 2: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.285 (0.166) | 0.377 (0.0531)
  Week 4: 0 hours: number analyzed (Participants) | 1 | 2 | 5 | 7
  Week 4: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.417 (0.143) | 0.414 (0.0742)
  Week 8: 0 hours: number analyzed (Participants) | 1 | 2 | 5 | 6
  Week 8: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.353 (0.226) | 0.466 (0.0913)
  Week 12: 0 hours: number analyzed (Participants) | 1 | 2 | 6 | 6
  Week 12: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.467 (0.188) | 0.479 (0.0650)
  Week 20: 0 hours: number analyzed (Participants) | 1 | 1 | 5 | 7
  Week 20: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.441 (0.147) | 0.481 (0.0625)
  Week 24: 0 hours: number analyzed (Participants) | 1 | 1 | 4 | 6
  Week 24: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.395 (0.309) | 0.385 (0.0415)
  Week 28: 0 hours: number analyzed (Participants) | 1 | 1 | 1 | 4
  Week 28: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.527 (0.0302)
  Week 32: 0 hours: number analyzed (Participants) | 1 | 0 | 1 | 4
  Week 32: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. |  | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.462 (0.0410)
  Week 36: 0 hours: number analyzed (Participants) | 1 | 0 | 1 | 4
  Week 36: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. |  | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.442 (0.0517)
  Week 44: 0 hours: number analyzed (Participants) | 1 | 0 | 1 | 3
  Week 44: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. |  | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.438 (0.0352)
  Week 48: 0 hours: number analyzed (Participants) | 1 | 0 | 3 | 4
  Week 48: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. |  | 0.434 (0.0968) | 0.539 (0.0414)
  Follow-up: Week 2: number analyzed (Participants) | 1 | 1 | 5 | 5
  Follow-up: Week 2 | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.542 (0.311) | 0.307 (0.176)
  Follow-up: Week 4: number analyzed (Participants) | 1 | 1 | 5 | 6
  Follow-up: Week 4 | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.354 (0.260) | 0.309 (0.161)

29. Secondary Outcome: Plasma Concentrations of ETV in Virologically Suppressed Population
Description: Plasma concentrations of ETV administered as monotherapy or co-administered with JNJ-56136379 in virologically suppressed population was determined. As planned, plasma concentration of ETV co-administered with placebo was analyzed separately for Part A and Part B. Samples were analyzed using POP PK modeling.
Time Frame: Day 1: 0 hours, 2 hours; Weeks 1, 2, 4, 8, 12, 20, 24, 28, 32, 36, 44, 48: 0 hours; Follow-up: Weeks 2 and 4
Population: The PK analysis set included data for all participants with available plasma concentrations. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) participants received matching placebo to JNJ-56136379 (75 milligrams [mg]) plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part B: Placebo (Matching to JNJ-56136379 250 mg) + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) participants received matching placebo to JNJ-56136379 (250 mg) plus 1 tablet of NA (05 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Virologically suppressed participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Virologically suppressed participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
Arm/Group | Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA) | Part B: Placebo (Matching to JNJ-56136379 250 mg) + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 4 | 2 | 14 | 6
ng/mL
  Day 1: 0 hours: number analyzed (Participants) | 1 | 0 | 7 | 0
  Day 1: 0 hours | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. |  | 0.683 (0.414) |
  Day 1: 2 hours: number analyzed (Participants) | 2 | 0 | 6 | 3
  Day 1: 2 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. |  | 1.86 (0.639) | 1.89 (0.429)
  Week 1: 0 hours: number analyzed (Participants) | 4 | 1 | 14 | 4
  Week 1: 0 hours | 1.94 (2.43) | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.464 (0.143) | 0.472 (0.120)
  Week 2: 0 hours: number analyzed (Participants) | 3 | 1 | 14 | 4
  Week 2: 0 hours | 0.871 (0.909) | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.469 (0.153) | 0.469 (0.0835)
  Week 4: 0 hours: number analyzed (Participants) | 3 | 1 | 10 | 4
  Week 4: 0 hours | 0.647 (0.628) | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.529 (0.198) | 0.539 (0.108)
  Week 8: 0 hours: number analyzed (Participants) | 2 | 1 | 11 | 4
  Week 8: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.496 (0.179) | 0.493 (0.0816)
  Week 12: 0 hours: number analyzed (Participants) | 3 | 1 | 11 | 4
  Week 12: 0 hours | 0.277 (0.0733) | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.454 (0.135) | 0.548 (0.0535)
  Week 20: 0 hours: number analyzed (Participants) | 2 | 1 | 10 | 4
  Week 20: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.617 (0.408) | 0.537 (0.109)
  Week 24: 0 hours: number analyzed (Participants) | 2 | 1 | 12 | 4
  Week 24: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | 0.491 (0.144) | 0.576 (0.121)
  Week 28: 0 hours: number analyzed (Participants) | 2 | 0 | 11 | 4
  Week 28: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. |  | 0.446 (0.148) | 0.519 (0.153)
  Week 32: 0 hours: number analyzed (Participants) | 2 | 0 | 11 | 4
  Week 32: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. |  | 0.467 (0.201) | 0.489 (0.144)
  Week 36: 0 hours: number analyzed (Participants) | 3 | 0 | 11 | 4
  Week 36: 0 hours | 0.962 (1.07) |  | 0.487 (0.185) | 0.526 (0.109)
  Week 44: 0 hours: number analyzed (Participants) | 2 | 0 | 11 | 4
  Week 44: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. |  | 0.525 (0.177) | 0.517 (0.121)
  Week 48: 0 hours: number analyzed (Participants) | 3 | 0 | 11 | 5
  Week 48: 0 hours | 0.766 (0.594) |  | 0.554 (0.287) | 0.537 (0.105)
  Follow-up: Week 2: number analyzed (Participants) | 2 | 2 | 11 | 6
  Follow-up: Week 2 | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.635 (0.449) | 0.433 (0.117)
  Follow-up: Week 4: number analyzed (Participants) | 3 | 2 | 10 | 6
  Follow-up: Week 4 | 1.00 (1.13) | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 0.445 (0.164) | 0.725 (0.598)

30. Secondary Outcome: Plasma Concentrations of Tenofovir Disoproxil Fumarate (TDF) in Currently Not Treated Population
Description: Plasma concentrations of TDF administered as monotherapy or co-administered with JNJ-56136379 was determined. As planned, plasma concentration of TDF co-administered with placebo was analyzed separately for Part A and Part B. Samples were analyzed using POP PK modeling.
Time Frame: Day 1: 0 hours, 2 hours; Weeks 1, 2, 4, 8, 12, 20, 24, 28, 32, 36, 44, 48: 0 hours; Follow-up: Weeks 2 and 4
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA): Currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (75 milligrams [mg]) plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part B: Placebo (Matching to JNJ-56136379 250 mg) + NA: Currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (250 mg) plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.)
Arm/Group | Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA) | Part B: Placebo (Matching to JNJ-56136379 250 mg) + NA | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 9 | 8 | 24 | 25
nanograms per milliliter (ng/mL)
  Day 1: 0 hours: number analyzed (Participants) | 2 | 1 | 4 | 4
  Day 1: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that mean and standard deviation was not estimable due to small sample size. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point.
  Day 1: 2 hours: number analyzed (Participants) | 9 | 7 | 22 | 25
  Day 1: 2 hours | 277 (116) | 170 (114) | 372 (478) | 249 (96.9)
  Week 1: 0 hours: number analyzed (Participants) | 9 | 8 | 24 | 24
  Week 1: 0 hours | 79.6 (38.1) | 92.7 (134) | 92.6 (37.4) | 97.8 (27.7)
  Week 2: 0 hours: number analyzed (Participants) | 9 | 8 | 22 | 24
  Week 2: 0 hours | 64.2 (34.5) | 50.1 (14.1) | 81.5 (22.6) | 97.6 (23.7)
  Week 4: 0 hours: number analyzed (Participants) | 9 | 7 | 22 | 24
  Week 4: 0 hours | 62.9 (17.7) | 46.5 (10.5) | 90.2 (25.8) | 99.6 (26.4)
  Week 8: 0 hours: number analyzed (Participants) | 9 | 7 | 23 | 23
  Week 8: 0 hours | 66.3 (23.7) | 54.2 (18.3) | 92.6 (25.7) | 108 (36.0)
  Week 12: 0 hours: number analyzed (Participants) | 9 | 7 | 24 | 23
  Week 12: 0 hours | 67.5 (31.2) | 51.3 (15.9) | 92.6 (29.1) | 102 (35.3)
  Week 20: 0 hours: number analyzed (Participants) | 9 | 7 | 24 | 23
  Week 20: 0 hours | 72.6 (34.2) | 51.2 (13.8) | 85.8 (30.6) | 115 (41.7)
  Week 24: 0 hours: number analyzed (Participants) | 9 | 7 | 23 | 23
  Week 24: 0 hours | 75.9 (51.0) | 50.5 (20.1) | 89.1 (30.1) | 99.3 (37.8)
  Week 28: 0 hours: number analyzed (Participants) | 6 | 5 | 9 | 17
  Week 28: 0 hours | 74.4 (38.1) | 51.2 (19.9) | 99.0 (32.6) | 108 (39.0)
  Week 32: 0 hours: number analyzed (Participants) | 6 | 5 | 8 | 16
  Week 32: 0 hours | 78.8 (59.6) | 52.7 (26.1) | 89.6 (37.1) | 88.5 (25.6)
  Week 36: 0 hours: number analyzed (Participants) | 5 | 5 | 9 | 16
  Week 36: 0 hours | 78.9 (55.8) | 42.5 (19.3) | 96.0 (38.3) | 101 (34.2)
  Week 44: 0 hours: number analyzed (Participants) | 6 | 5 | 8 | 16
  Week 44: 0 hours | 86.3 (30.8) | 46.3 (26.0) | 81.8 (38.9) | 105 (33.5)
  Week 48: 0 hours: number analyzed (Participants) | 6 | 4 | 8 | 15
  Week 48: 0 hours | 76.4 (40) | 47.8 (18.6) | 89.5 (49.8) | 100 (29.9)
  Follow-up: Week 2: number analyzed (Participants) | 8 | 7 | 21 | 19
  Follow-up: Week 2 | 73.8 (37.1) | 52.1 (17.3) | 65.7 (29.5) | 73.5 (23.2)
  Follow-up: Week 4: number analyzed (Participants) | 9 | 7 | 22 | 21
  Follow-up: Week 4 | 72.4 (32.1) | 57.1 (13.6) | 68.7 (54.3) | 68.4 (43.6)

31. Secondary Outcome: Plasma Concentrations of TDF in Virologically Suppressed Population
Description: as for outcome 30
Time Frame: Day 1: 0 hours, 2 hours; Weeks 1, 2, 4, 8, 12, 20, 24, 28, 32, 36, 44, 48: 0 hours; Follow-up: Weeks 2 and 4
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) participants received matching placebo to JNJ-56136379 (75 milligrams [mg]) plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part B: Placebo (Matching JNJ-56136379 250 mg) + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) participants received matching placebo to JNJ-56136379 (250 mg) plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA: Virologically suppressed participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA: Virologically suppressed participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
Arm/Group | Part A: Placebo (Matching JNJ-56136379 75 mg) + Nucleos(t)Ide Analog (NA) | Part B: Placebo (Matching JNJ-56136379 250 mg) + Nucleos(t)Ide Analog (NA) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 5 | 8 | 18 | 19
ng/mL
  Day 1: 0 hours: number analyzed (Participants) | 2 | 2 | 3 | 4
  Day 1: 0 hours | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 68.9 (10.1) | 63.3 (27.4)
  Day 1: 2 hours: number analyzed (Participants) | 3 | 8 | 18 | 16
  Day 1: 2 hours | 274 (153) | 311 (92.5) | 306 (145) | 364 (260)
  Week 1: 0 hours: number analyzed (Participants) | 5 | 8 | 18 | 18
  Week 1: 0 hours | 76.8 (40.8) | 59.2 (15.7) | 97.9 (38.0) | 97.1 (36.8)
  Week 2: 0 hours | 82.0 (53.0) | 65.9 (18.9) | 97.5 (34.0) | 114 (51.0)
  Week 4: 0 hours: number analyzed (Participants) | 5 | 6 | 18 | 18
  Week 4: 0 hours | 83.1 (54.8) | 66.9 (20.3) | 96.9 (25.0) | 110 (41.4)
  Week 8: 0 hours: number analyzed (Participants) | 4 | 7 | 18 | 19
  Week 8: 0 hours | 84.0 (54.1) | 65.5 (28.9) | 118 (48.0) | 109 (32.2)
  Week 12: 0 hours: number analyzed (Participants) | 4 | 7 | 18 | 18
  Week 12: 0 hours | 98.8 (73.6) | 63.5 (21.6) | 99.4 (33.8) | 130 (87.8)
  Week 20: 0 hours: number analyzed (Participants) | 4 | 7 | 15 | 18
  Week 20: 0 hours | 99.6 (85.0) | 64.8 (23.3) | 120 (30.1) | 127 (64.9)
  Week 24: 0 hours: number analyzed (Participants) | 5 | 7 | 15 | 16
  Week 24: 0 hours | 78.3 (33.4) | 73.8 (33.0) | 104 (29.9) | 113 (47.6)
  Week 28: 0 hours: number analyzed (Participants) | 4 | 6 | 14 | 16
  Week 28: 0 hours | 81.7 (37.7) | 70.6 (28.1) | 110 (43.2) | 155 (107)
  Week 32: 0 hours: number analyzed (Participants) | 5 | 6 | 13 | 14
  Week 32: 0 hours | 75.5 (54.8) | 61.2 (21.2) | 43.2 (36.4) | 139 (93.3)
  Week 36: 0 hours: number analyzed (Participants) | 5 | 6 | 14 | 14
  Week 36: 0 hours | 80.2 (50.3) | 80.2 (31.2) | 101 (33.1) | 132 (90.2)
  Week 44: 0 hours: number analyzed (Participants) | 5 | 6 | 13 | 11
  Week 44: 0 hours | 72.7 (54.9) | 93.0 (64.2) | 109 (53.4) | 129 (73.6)
  Week 48: 0 hours: number analyzed (Participants) | 5 | 6 | 13 | 10
  Week 48: 0 hours | 87.6 (58.5) | 66.2 (22.1) | 114 (31.7) | 133 (117)
  Follow-up: Week 2: number analyzed (Participants) | 4 | 6 | 12 | 10
  Follow-up: Week 2 | 86.5 (73.8) | 51.9 (23.4) | 73.2 (18.5) | 136 (95.5)
  Follow-up: Week 4: number analyzed (Participants) | 5 | 7 | 14 | 9
  Follow-up: Week 4 | 74.7 (47.6) | 59.7 (23.4) | 71.2 (33.0) | 95.8 (83.6)

32. Secondary Outcome: Plasma Concentrations of JNJ-56136379 in Currently Not Treated Population
Description: Plasma concentrations of JNJ-56136379 in currently not treated population administered as monotherapy or when co-administered with NA (ETV or TDF) was determined. As planned, the plasma concentration of JNJ-56136379 when co-administered with NA was determined separately for each NA treatment (ETV and TDF). Samples were analyzed using POP PK modeling.
Time Frame: Day 1: 0 hours, 2 hours; Weeks 1, 2, 4, 8, 12, 20, 24, 28, 32, 36, 44, 48: 0 hours; Follow-up: Weeks 2 and 4
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part A: JNJ-56136379 75 mg (Open Label): Currently not treated participants received 3*25 mg tablets of JNJ-56136379 once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued treatment with JNJ-56136379 75 mg from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and receive treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA (ETV): Currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA (TDF): Currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA (ETV): Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA (TDF): Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
Arm/Group | Part A: JNJ-56136379 75 mg (Open Label) | Part B: JNJ-56136379 250 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA (ETV) | Part A: JNJ-56136379 75 mg + NA (TDF) | Part B: JNJ-56136379 250 mg + NA (ETV) | Part B: JNJ-56136379 250 mg + NA (TDF)
Number analyzed (Participants) | 27 | 32 | 8 | 24 | 7 | 25
ng/mL
  Day 1: 0 hour: number analyzed (Participants) | 6 | 4 | 2 | 4 | 3 | 4
  Day 1: 0 hour | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due to below qualification limit (BQL) that is <10.0 ng/mL. | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due to below qualification limit (BQL) that is <10.0 ng/mL. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due to below qualification limit (BQL) that is <10.0 ng/mL. | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due below qualification limit BQL limit <10.0 ng/mL. | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due below qualification limit BQL limit <10.0 ng/mL.
  Day 1: 2 hour: number analyzed (Participants) | 24 | 27 | 8 | 22 | 6 | 25
  Day 1: 2 hour | 709 (307) | 2143 (1300) | 520 (279) | 806 (306) | 2287 (946) | 2021 (893)
  Week 1: 0 hours: number analyzed (Participants) | 27 | 30 | 8 | 24 | 7 | 24
  Week 1: 0 hours | 2269 (597) | 7339 (2040) | 2264 (455) | 2368 (695) | 6461 (2014) | 7138 (2280)
  Week 2: 0 hours: number analyzed (Participants) | 26 | 31 | 8 | 23 | 7 | 24
  Week 2: 0 hours | 3424 (845) | 10894 (2631) | 3094 (892) | 3702 (1028) | 9381 (2168) | 10588 (3568)
  Week 4: 0 hours: number analyzed (Participants) | 27 | 31 | 8 | 23 | 7 | 24
  Week 4: 0 hours | 4116 (941) | 12827 (3104) | 4368 (1216) | 4697 (1474) | 10760 (2162) | 12513 (4229)
  Week 8: 0 hours: number analyzed (Participants) | 26 | 31 | 8 | 24 | 7 | 22
  Week 8: 0 hours | 4617 (1195) | 13697 (3702) | 5006 (1528) | 4719 (1465) | 11027 (2009) | 13037 (4394)
  Week 12: 0 hours: number analyzed (Participants) | 26 | 29 | 8 | 24 | 7 | 23
  Week 12: 0 hours | 4130 (1145) | 12676 (3431) | 4976 (1302) | 4582 (1324) | 11347 (1754) | 12524 (4756)
  Week 20: 0 hours: number analyzed (Participants) | 22 | 30 | 8 | 24 | 7 | 23
  Week 20: 0 hours | 3754 (1132) | 12757 (4298) | 4648 (1528) | 4698 (1661) | 10517 (2031) | 11425 (3719)
  Week 24: 0 hours: number analyzed (Participants) | 8 | 21 | 3 | 14 | 4 | 21
  Week 24: 0 hours | 3613 (813) | 12626 (3396) | 4650 (1461) | 4767 (1601) | 10888 (1576) | 11625 (5087)
  Week 28: 0 hours: number analyzed (Participants) | 3 | 20 | 3 | 9 | 4 | 17
  Week 28: 0 hours | 4733 (350) | 12025 (3229) | 4300 (1355) | 4439 (1446) | 11753 (2719) | 11746 (4752)
  Week 32: 0 hours: number analyzed (Participants) | 0 | 20 | 3 | 8 | 4 | 17
  Week 32: 0 hours |  | 12162 (2780) | 4677 (646) | 4825 (2429) | 9840 (3770) | 12119 (4062)
  Week 36: 0 hours: number analyzed (Participants) | 0 | 19 | 3 | 9 | 4 | 17
  Week 36: 0 hours |  | 11289 (2973) | 4463 (1444) | 4144 (1599) | 11350 (3439) | 11192 (5191)
  Week 44: 0 hours: number analyzed (Participants) | 0 | 9 | 3 | 8 | 4 | 17
  Week 44: 0 hours |  | 11198 (2749) | 4507 (1121) | 3430 (1346) | 11570 (2674) | 11016 (4277)
  Week 48: 0 hours: number analyzed (Participants) | 0 | 32 | 0 | 2 | 3 | 10
  Week 48: 0 hours |  | 11797 (2482) |  | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 11220 (2464) | 10740 (2400)
  Follow-up: Week 2: number analyzed (Participants) | 21 | 28 | 8 | 21 | 7 | 19
  Follow-up: Week 2 | 916 (930) | 2459 (1529) | 1330 (887) | 909 (740) | 1922 (1628) | 2192 (1535)
  Follow-up: Week 4: number analyzed (Participants) | 22 | 29 | 8 | 22 | 6 | 21
  Follow-up: Week 4 | 242 (359) | 494 (427) | 320 (276) | 226 (236) | 572 (624) | 1025 (1523)

33. Secondary Outcome: Plasma Concentrations of JNJ-56136379 in Virologically Suppressed Population
Description: Plasma concentrations of JNJ-56136379 in virologically suppressed population administered as monotherapy or when co-administered with NA (ETV or TDF) was determined. As planned, the plasma concentration of JNJ-56136379 when co-administered with NA was determined separately for each NA treatment (ETV and TDF). Samples were analyzed using POP PK modeling.
Time Frame: Day 1: 0 hours, 2 hours; Weeks 1, 2, 4, 8, 12, 20, 24, 28, 32, 36, 44, 48: 0 hours; Follow-up: Weeks 2 and 4
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part A: JNJ-56136379 75 mg + NA (ETV): Virologically suppressed participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part A: JNJ-56136379 75 mg + NA (TDF): Virologically suppressed participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA (ETV): Virologically suppressed participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (0.5 mg ETV) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (ETV) for additional 24 weeks.
- Part B: JNJ-56136379 250 mg + NA (TDF): Virologically suppressed participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA (300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who did not participate in the treatment extension phase after Week 24 and those who completed the extension phase were followed up and continued treatment with only NA (TDF) for additional 24 weeks.
Arm/Group | Part A: JNJ-56136379 75 mg + NA (ETV) | Part A: JNJ-56136379 75 mg + NA (TDF) | Part B: JNJ-56136379 250 mg + NA (ETV) | Part B: JNJ-56136379 250 mg + NA (TDF)
Number analyzed (Participants) | 15 | 17 | 8 | 19
ng/mL
  Day 1: 0 hour: number analyzed (Participants) | 6 | 2 | 0 | 4
  Day 1: 0 hour | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due to below qualification limit (BQL) that is <10.0 ng/mL. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. |  | NA (NA) — Here "NA" indicates that mean and standard deviation was not calculated due to below qualification limit (BQL) that is <10.0 ng/mL.
  Day 1: 2 hour: number analyzed (Participants) | 13 | 16 | 7 | 17
  Day 1: 2 hour | 857 (238) | 616 (385) | 2103 (1400) | 2083 (1022)
  Week 1: 0 hours: number analyzed (Participants) | 15 | 16 | 8 | 18
  Week 1: 0 hours | 2144 (553) | 2301 (639) | 5758 (1081) | 7280 (2098)
  Week 2: 0 hours | 3193 (1017) | 3206 (710) | 8485 (2269) | 10077 (2886)
  Week 4: 0 hours: number analyzed (Participants) | 15 | 16 | 8 | 19
  Week 4: 0 hours | 3689 (1178) | 3694 (815) | 10106 (2838) | 12167 (4271)
  Week 8: 0 hours | 3917 (1131) | 3998 (1376) | 11295 (3829) | 13352 (6072)
  Week 12: 0 hours: number analyzed (Participants) | 14 | 16 | 8 | 18
  Week 12: 0 hours | 4194 (1279) | 3813 (945) | 10404 (4246) | 12776 (5191)
  Week 20: 0 hours: number analyzed (Participants) | 15 | 17 | 8 | 18
  Week 20: 0 hours | 3948 (1151) | 4134 (1375) | 10761 (3980) | 12432 (4249)
  Week 24: 0 hours: number analyzed (Participants) | 14 | 17 | 8 | 16
  Week 24: 0 hours | 3989 (957) | 3836 (1160) | 10219 (3370) | 11542 (4612)
  Week 28: 0 hours: number analyzed (Participants) | 15 | 16 | 8 | 16
  Week 28: 0 hours | 4259 (1083) | 3506 (1032) | 9959 (2929) | 11344 (4482)
  Week 32: 0 hours: number analyzed (Participants) | 15 | 14 | 8 | 14
  Week 32: 0 hours | 3788 (841) | 3721 (1088) | 10189 (3160) | 12099 (6301)
  Week 36: 0 hours: number analyzed (Participants) | 15 | 15 | 8 | 14
  Week 36: 0 hours | 3801 (1170) | 3535 (964) | 10036 (2786) | 12227 (5396)
  Week 44: 0 hours: number analyzed (Participants) | 15 | 14 | 8 | 12
  Week 44: 0 hours | 3998 (1139) | 3784 (1056) | 9634 (3707) | 14853 (7977)
  Week 48: 0 hours: number analyzed (Participants) | 5 | 2 | 2 | 6
  Week 48: 0 hours | 3918 (1259) | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | NA (NA) — Here "NA" indicates that actual sampling time deviated too much from nominal scheduled sampling time. Therefore, data could not be estimated and analyzed at specific time point. | 15080 (8060)
  Follow-up: Week 2: number analyzed (Participants) | 14 | 13 | 8 | 14
  Follow-up: Week 2 | 621 (607) | 912 (585) | 1919 (1359) | 3190 (4462)
  Follow-up: Week 4: number analyzed (Participants) | 15 | 14 | 8 | 15
  Follow-up: Week 4 | 89.8 (102) | 204 (209) | 389 (384) | 1066 (2319)

34. Secondary Outcome: Number of Participants With Treatment-Associated Mutations
Description: Number of participants with treatment-associated mutations were reported. Viral genome sequence analysis was performed to evaluate emergence of mutations associated with JNJ-56136379 considering 15 HBV core protein positions of interest. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: From Week 0 to Week 24, From Week 25 to Week 48, Up to Follow-up Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: JNJ-56136379 75 mg (Open Label) | Part A: JNJ-56136379 75 mg + NA | Part B: JNJ-56136379 250 mg (Open Label) | Part B: JNJ-56136379 250 mg + NA
Number analyzed (Participants) | 23 | 22 | 17 | 14
Participants
  Emergence of mutations during 24 weeks (Week 0 to Week 24) | 8 | 0 | 4 | 0
  Emergence of mutations between 25 and 48 weeks (Week 25 to Week 48) | 2 | 0 | 0 | 0
  Emergence of mutations on NA treatment (Up to Follow-up Week 24) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening to end of study (up to Week 80) (Screening period of 8 weeks + Initial treatment phase of 24 weeks [Week 0 to Week 24] + 24 week Follow-up [Week 0 to Week 48], and Treatment extension phase of 24 weeks [Week 24 to Week 48] + 24 week follow-up [Week 24 to Week 72]= Week 80)
Description: Safety analysis set included all participants who received at least one dose of the study agent and all safety endpoints analyzed by the treatment arm as treated.
Groups:
- Initial Treatment Phase: Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA): Virologically suppressed (who were on entecavir [ETV] or tenofovir disoproxil fumarate [TDF] for at least 12 months prior to screening and had hepatitis B virus [HBV] deoxyribonucleic acid [DNA] <60 IU/ml) or currently not treated (who didn't receive any HBV treatment 6 months prior to baseline) participants received matching placebo to JNJ-56136379 (75 milligrams [mg] or 250 mg) plus 1 tablet of NA (either 0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who did not participate in the treatment extension phase after Week 24 were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Initial Treatment Phase: Part A: JNJ-56136379 75 mg (Open Label): Currently not treated participants received 3*25 mg tablets of JNJ-56136379 once daily from Day 1 to Week 24 during the initial treatment phase. Participants who did not participate in the treatment extension phase after Week 24 were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Initial Treatment Phase: Part A: JNJ-56136379 75 mg + NA: Virologically suppressed or currently not treated participants received 3*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during the initial treatment phase. Participants who did not participate in the treatment extension phase after Week 24 were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Initial Treatment Phase: Part B: JNJ-56136379 250 mg (Open-label): Currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 once daily from Day 1 to Week 24 during the initial treatment phase. Participants who did not participate in the treatment extension phase after Week 24 were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Initial Treatment Phase: Part B: JNJ-56136379 250 mg + NA: Virologically suppressed or currently not treated participants received 2*100 mg and 2*25 mg tablets of JNJ-56136379 plus 1 tablet of NA either (0.5 mg ETV or 300 mg TDF) once daily from Day 1 to Week 24 during treatment phase. Participants who did not participate in the treatment extension phase after Week 24 were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Treatment Extension Phase: Parts A and B: Pooled Placebo + NA: Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Treatment Extension Phase: Part A: JNJ-56136379 75 mg (Open Label): Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued treatment with JNJ-56136379 75mg from Week 24 to Week 48 in the treatment extension phase. Participants who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Treatment Extension Phase: Part A: JNJ-56136379 75 mg + NA: Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 75 mg treatment from Week 24 to Week 48 in the treatment extension phase. Participants who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Treatment Extension Phase: Part B: JNJ-56136379 250 mg (Open-label): Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants who completed the extension phase were followed up and received treatment with only NA (either ETV or TDF) for additional 24 weeks.
- Treatment Extension Phase: Part B: JNJ-56136379 250 mg + NA: Participants who completed the initial 24 weeks of treatment with a virologic response by Week 20 and without experiencing any safety concerns precluding continued JNJ-56136379 treatment from Week 24 to Week 48 in the treatment extension phase. Participants those who completed the extension phase were followed up and continued treatment with only NA (either ETV or TDF) for additional 24 weeks.
Arm/Group | Initial Treatment Phase: Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) | Initial Treatment Phase: Part A: JNJ-56136379 75 mg (Open Label) | Initial Treatment Phase: Part A: JNJ-56136379 75 mg + NA | Initial Treatment Phase: Part B: JNJ-56136379 250 mg (Open-label) | Initial Treatment Phase: Part B: JNJ-56136379 250 mg + NA | Treatment Extension Phase: Parts A and B: Pooled Placebo + NA | Treatment Extension Phase: Part A: JNJ-56136379 75 mg (Open Label) | Treatment Extension Phase: Part A: JNJ-56136379 75 mg + NA | Treatment Extension Phase: Part B: JNJ-56136379 250 mg (Open-label) | Treatment Extension Phase: Part B: JNJ-56136379 250 mg + NA
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/28 | 0/66 | 0/32 | 0/63 | 0/33 | 0/3 | 0/43 | 0/20 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/28 | 0/66 | 0/32 | 1/63 | 0/33 | 0/3 | 4/43 | 0/20 | 3/48
Other Adverse Events (participants affected / at risk) | 9/43 | 18/28 | 19/66 | 12/32 | 11/63 | 25/33 | 2/3 | 38/43 | 15/20 | 42/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Phase: Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) (N=43) | Initial Treatment Phase: Part A: JNJ-56136379 75 mg (Open Label) (N=28) | Initial Treatment Phase: Part A: JNJ-56136379 75 mg + NA (N=66) | Initial Treatment Phase: Part B: JNJ-56136379 250 mg (Open-label) (N=32) | Initial Treatment Phase: Part B: JNJ-56136379 250 mg + NA (N=63) | Treatment Extension Phase: Parts A and B: Pooled Placebo + NA (N=33) | Treatment Extension Phase: Part A: JNJ-56136379 75 mg (Open Label) (N=3) | Treatment Extension Phase: Part A: JNJ-56136379 75 mg + NA (N=43) | Treatment Extension Phase: Part B: JNJ-56136379 250 mg (Open-label) (N=20) | Treatment Extension Phase: Part B: JNJ-56136379 250 mg + NA (N=48)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Failure Acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toxic Shock Syndrome Streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Initial Treatment Phase: Parts A and B: Pooled Placebo + Nucleos(t)Ide Analog (NA) (N=43) | Initial Treatment Phase: Part A: JNJ-56136379 75 mg (Open Label) (N=28) | Initial Treatment Phase: Part A: JNJ-56136379 75 mg + NA (N=66) | Initial Treatment Phase: Part B: JNJ-56136379 250 mg (Open-label) (N=32) | Initial Treatment Phase: Part B: JNJ-56136379 250 mg + NA (N=63) | Treatment Extension Phase: Parts A and B: Pooled Placebo + NA (N=33) | Treatment Extension Phase: Part A: JNJ-56136379 75 mg (Open Label) (N=3) | Treatment Extension Phase: Part A: JNJ-56136379 75 mg + NA (N=43) | Treatment Extension Phase: Part B: JNJ-56136379 250 mg (Open-label) (N=20) | Treatment Extension Phase: Part B: JNJ-56136379 250 mg + NA (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Defect Conduction Intraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ear Congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Motion Sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling of Eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 4
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 3 | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faeces Hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 2 | 3 | 0 | 1 | 1 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 4 | 1 | 1 | 4 | 0 | 4 | 1 | 4
Influenza Like Illness (General disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Pain (Hepatobiliary disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular Icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alveolar Osteitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Bronchitis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helicobacter Gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 3 | 2 | 7 | 0 | 5 | 1 | 8
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 1
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulpitis Dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Suspected Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 8 | 4 | 4
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Vulvitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 3 | 4
Amylase Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Calcium Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 3 | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood Glucose Increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Magnesium Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood Potassium Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Triglycerides (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram T Wave Inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis B Dna Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Protein Urine Present (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sars-Cov-2 Test Positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ultrasound Liver Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Sediment Present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine Analysis Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine Leukocyte Esterase Positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 5 | 2 | 3
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint Noise (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0/23 | 0 | 0 | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 5 | 3 | 2 | 4 | 0 | 6 | 4 | 12
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuromuscular Pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parkinson's Disease (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor Quality Sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Discomfort (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 3
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Alopecia Areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 2
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abortion Induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental Implantation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03361956/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03361956/SAP_001.pdf